CLINICAL TRIAL: NCT06692790
Title: Venous StEnt for Idiopathic IntraCranial HypertEnsion (VEHICLE) Registry: Management and Outcomes in the MENA Region
Brief Title: VEHICLE Registry: Venous Stenting for IIH in the MENA Region
Acronym: VEHICLE
Status: Recruiting | Type: Observational
Sponsor: Middle East North Africa Stroke and Interventional Neurotherapies Organization (Other)
Responsible Party: Principal Investigator, Ossama Mansour, Professor of Neurology and stroke, Middle East North Africa Stroke and Interventional Neurotherapies Organization
Other Study IDs: MENASINO1001S
Record Dates: First submitted 2024-11-15; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-05

CONDITIONS: Idiopathic Intracranial Hypertension (IIH)
Keywords: Venous Sinus Stenosis; Venous Sinus Stenting; Papilledema; Middle East and North Africa (MENA); Magnetic Resonance Venography (MRV)
MeSH Terms: conditions — Pseudotumor Cerebri; Papilledema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Venous Sinus Stenting Procedure — Performed under general or local anesthesia. Targeted stenosis sites included the right transverse sinus, left transverse sinus, bilateral transverse sinuses, and right transverse and sigmoid sinuses.
  Stents used included Venous Sinus Stent (CWS), CASPER, PRTCS, and multiple stents where necessary.
  Post-procedure care included antiplatelet therapy and routine follow-up assessments

SUMMARY:
The VEHICLE Registry is a multicenter observational study aimed at evaluating the management and outcomes of patients with Idiopathic Intracranial Hypertension (IIH) undergoing venous sinus stenting in the Middle East and North Africa (MENA) region. The study focuses on assessing clinical characteristics, treatment efficacy, safety, and the role of venous sinus stenting as a therapeutic modality in IIH.

DETAILED DESCRIPTION:
Idiopathic Intracranial Hypertension (IIH) is a condition characterized by elevated intracranial pressure without an identifiable cause, leading to symptoms such as headaches, visual disturbances, and potential vision loss due to papilledema. The condition predominantly affects obese women of childbearing age and is associated with risk factors like obesity, recent weight gain, hypothyroidism, and polycystic ovary syndrome (PCOS).

Venous sinus stenosis has been implicated in the pathophysiology of IIH. Venous sinus stenting has emerged as a promising treatment option for patients who are refractory to medical therapy or intolerant to medications like acetazolamide.

The VEHICLE Registry collects real-world data from multiple centers in the MENA region to evaluate the efficacy and safety of venous sinus stenting in patients with IIH. The registry analyzes patient demographics, clinical presentations, imaging findings, treatment details, and outcomes over a six-month follow-up period to improve understanding and management of IIH in this population.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 60 years.

Diagnosed with Idiopathic Intracranial Hypertension (IIH) based on the modified Dandy criteria, including:

Symptoms of increased intracranial pressure (e.g., headache, visual disturbances).

Elevated opening pressure (>250 mm H₂O) on lumbar puncture with normal cerebrospinal fluid composition.

No evidence of intracranial pathology (e.g., mass lesion, hydrocephalus) on neuroimaging.

Presence of papilledema. Evidence of venous sinus stenosis on Magnetic Resonance Venography (MRV) or Digital Subtraction Angiography (DSA).

Refractory to medical therapy or intolerant to medications (e.g., acetazolamide).

Willingness to undergo venous sinus stenting. Provided informed consent for participation.

Exclusion Criteria:

* Secondary causes of intracranial hypertension (e.g., cerebral venous sinus thrombosis, neoplasm).

Coagulopathies or contraindications to antiplatelet or anticoagulation therapy. Pregnancy or lactation. Incomplete baseline data or inability to complete follow-up assessments. Severe comorbid conditions that preclude endovascular procedures.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients diagnosed with Idiopathic Intracranial Hypertension who are candidates for venous sinus stenting, recruited from multiple centers across the MENA region.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-08-11 (Actual); Primary Completion 2025-08-11 (Estimated); Study Completion 2025-11-11 (Estimated)

PRIMARY OUTCOMES:
Symptom Improvement | Six months post-procedure.
  Proportion of patients reporting significant improvement or resolution of IIH symptoms (headache, visual disturbances, tinnitus) at six months post-venous sinus stenting.
Change in Papilledema Grade | Six months post-procedure.
  Improvement in papilledema grade assessed by fundoscopic examination using the Frisén scale from baseline to six months post-procedure.
Quality of Life Improvement | Baseline and six months post-procedure.
  Change in Quality of Life (QOL) scores measured using a standardized questionnaire from baseline to six months post-procedure.

SECONDARY OUTCOMES:
Stent Patency Rate | Six months post-procedure.
  Proportion of patients with patent venous sinus stents as assessed by imaging (MRV or DSA) at six months follow-up.
Adverse Events | Up to six months post-procedure.
  Incidence of procedural complications or adverse events related to venous sinus stenting within six months post-procedure.
Visual Field Improvement | Six months post-procedure.
  Improvement in visual field defects assessed by perimetry testing at six months post-procedure.
Cranial Neuropathy Resolution | Six months post-procedure.
  Resolution or improvement of cranial neuropathies (e.g., sixth nerve palsy) at six months post-procedure.

CONTACTS AND LOCATIONS:
Locations (2):
- Alexandria University, Alexandria, Egypt
- King Abdullah Medical City (KAMC) -, Mecca, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
The VEHICLE Registry plans to share de-identified individual participant data (IPD) to promote transparency and facilitate further research in the field of Idiopathic Intracranial Hypertension (IIH). Sharing this data aims to contribute to a better understanding of IIH management and outcomes, especially regarding venous sinus stenting in the Middle East and North Africa (MENA) region.
Supporting Information: Study Protocol
Time Frame: Data will be available beginning 6 months after publication of the primary study results.
  Data availability will continue for a period of 5 years following the initial publication.
Access Criteria: Qualified researchers affiliated with academic institutions, research organizations, or medical institutions.
  Researchers who provide a methodologically sound research proposal that is approved by an independent review committee.